CLINICAL TRIAL: NCT01201369
Title: Comparison of Rates of Strut Malapposition Between Everolimus and Sirolimus Eluting Stents - A Randomised Optical Coherence Tomography Study
Brief Title: A Study to Examine the Implantation Characteristics of Two Drug-Eluting Stents
Acronym: ORCA-2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Royal Brompton & Harefield NHS Foundation Trust (Other)
Responsible Party: Dr Miles Dalby, Consultant Cardiologist, Royal Brompton & Harefield NHS Foundation Trust
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ORCA-2
Record Dates: First submitted 2010-08-24; First posted 2010-09-14 (Estimated); Last update posted 2011-07-12 (Estimated); Status verified 2011-07

CONDITIONS: Coronary Artery Disease
Keywords: Percutaneous Coronary Intervention; Coronary Artery Stenosis; Acute Myocardial Infarction; Coronary Artery Stent; Optical Coherence Tomography
MeSH Terms: conditions — Coronary Artery Disease; Coronary Stenosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cypher™ Stent (Active Comparator): Participants in the Cypher arm will be randomised to receive a Cypher™ (Cordis, Miami Lake, USA) coronary stent
  Interventions: Device: Coronary Stent Cypher
- Xience™ Stent (Active Comparator): Patients in the Xience™ arm will receive a Xience™ Stent(Abbott Vascular, Santa Clara, USA.
  Interventions: Device: Coronary stent Xience

INTERVENTIONS:
Device: Coronary Stent Cypher — The angioplasty will then be performed in a usual fashion in accordance with the operator's discretion and local protocols.
  Arms: Cypher™ Stent
Device: Coronary stent Xience — The angioplasty will then be performed in a usual fashion in accordance with the operator's discretion and local protocols
  Arms: Xience™ Stent

SUMMARY:
Despite recent advances in stent technology and clot reducing drug therapy, acute stent occlusion or thrombosis (ST), still occurs and can be life threatening. It has been shown that certain features of how the stent relates to the artery wall may predict ST. One such feature, so-called stent strut malapposition (SSM), can be assessed after implantation but current imaging techniques are relatively unreliable. Optical Coherence Tomography (OCT) is a newer technology that can be performed safely and easily after angioplasty and may allow the stent struts to be assessed more accurately and reliably.

This study will use OCT to examine how two different types of commonly used drug-eluting stents relate to the artery wall. The Xience V (Abbott Vascular, USA) stent has thinner struts and a more open frame than the Cypher (Cordis, USA) stent. We hypothesise therefore that the potentially more pliable structure of the Xience V stent will be associated with greater contact with the vessel wall. This may have a bearing on the relative rate of SSM, although large studies have shown the rate to be low in both the Cypher and the Xience V stent. We believe that OCT imaging of SSM and symmetry of the stent immediately after angioplasty will compliment conventional visual assessment and may identify those patients in whom further improvement of stent with a balloon is necessary.

This study will involve the random allocation of forty patients requiring coronary angioplasty to one of the Cypher or Xience V stent. The procedure will be performed in the usual manner as indicated clinically and will include imaging of the stented artery segment with OCT once the operator is satisfied with the visual result by angiography.

ELIGIBILITY:
Inclusion Criteria:

* Presence of a coronary artery stenosis undergoing percutaneous coronary intervention and stenting (PCI).
* Eligibility for drug eluting stent (DES) deployment.
* Stable or unstable coronary syndrome presentation, including ST elevation myocardial infarction (STEMI).
* Aged 18-90

Exclusion Criteria:

* Contraindication to the use of a DES.
* Target lesion located within previous stent (in stent restenosis).
* Sustained haemodynamic instability following stent deployment (Systolic BP 90≤ mmHg or sustained ventricular arrhythmia).

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2010-09; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
Stent strut malapposition (SSM) | Immediate post stent deployment during the same angiographic procedure within 60 minutes
  SSM will be quoted as the percentage of malapposed stent struts as a proportion of the total number of struts analysed within each stent group.

SECONDARY OUTCOMES:
Stent eccentricity index (SEI) | Immediate post stent deployment during the same angiographic procedure within 60 minutes
  This is a commonly used measure that is designed to quantify the uniformity and symmetry of the stent after it has been deployed in the coronary artery. It is calculated as the minimum diameter of the stent divided by the maximum diameter of the stent at a preset point. The mean SEI will be compared between two stent type groups.
Degree of stent embedding | Immediate post stent deployment during the same angiographic procedure within 60 minutes
  This relates to what degree, if at all, the stent strut is 'buried' within the coronary artery wall. The proportion of each strut that is buried or embedded will be calculated and then averaged for each stent group. A strut that is buried in the vessel wall for more than half its thickness will be defined as 'embedded'.

CONTACTS AND LOCATIONS:
Overall Officials: Miles CD Dalby, MD, MRCP, Principal Investigator — Consultant Cardiologist, The Royal Brompton & Harefield NHS Foundation Trust; Robert D Smith, MD, MRCP, Study Director — The Royal Brompton & Harefield NHS Foundation Trust
Locations (1):
- Harefield Hospital, Harefield, Middlesex, United Kingdom